CLINICAL TRIAL: NCT05840991
Title: Effect of Short-term Compression Therapy After Thermal Ablation for Varicose Veins : a Prospective, Multicenter, Non-inferiority, Randomized Controlled Trial
Brief Title: Effect of Short-term Compression Therapy After Thermal Ablation for Varicose Veins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); China-Japan Union Hospital, Jilin University (Other); Yantai Yuhuangding Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Affiliated Hospital of Shaoxing University (Unknown); Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K2023047
Record Dates: First submitted 2023-04-17; First posted 2023-05-03 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Varicose Veins
Keywords: Varicose veins; Thermal ablation; Compression therapy; Targeted vein occlusion rate; Randomized controlled trial
MeSH Terms: conditions — Varicose Veins | interventions — Compression Bandages; Stockings, Compression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term compression group (Experimental): Patients randomised to group A will be provided with bandages to wear for 48 hours only
  Interventions: Device: elastic bandage
- Long-term compression group (Active Comparator): Patients randomised to group B will be asked to wear bandages for the first 24h and then a Class 2 compression full-length stocking (23-32mm Hg) for 1 week
  Interventions: Device: elastic bandage; Device: compression stocking

INTERVENTIONS:
Device: elastic bandage — 3M™ Coban™ elastic bandage
Device: compression stocking — Class 2 compression full-length stocking (23-32mm Hg)
  Arms: Long-term compression group

SUMMARY:
A prospective, multicenter, non-inferiority, randomized controlled trial is designed to evaluate the effect after short-term compression therapy following thermal ablation of varicose veins. Patients will be randomly assigned in a 1:1 ratio to one of the following treatments: (A) elastic bandage for 48h or (B) elastic bandage for the first 24h and then a compression full-length stocking (23-32mm Hg) for 1 week. The two groups will be compared on several variables, including target vein occlusion rate at 3 months (primary outcome indicator) , as well as pain, quality of life, clinical severity of varicose veins, postoperative complications, time to return to normal work, and compliance.

DETAILED DESCRIPTION:
A prospective, multicenter, non-inferiority, randomized controlled trial is designed to evaluate the effect after short-term compression therapy following thermal ablation of varicose veins. Patients will be randomly assigned in a 1:1 ratio to one of the following treatments: (A) elastic bandage for 48h or (B) elastic bandage for the first 24h and then a compression full-length stocking (23-32mm Hg) for 1 week. The two groups will be compared on several variables, including target vein occlusion rate at 3 months (primary outcome indicator) , as well as pain, quality of life, clinical severity of varicose veins, postoperative complications, time to return to normal work, and compliance.

The current study will take place in nine hospitals in six provinces in China. Target Population Patients referred to those with primary lower extremity saphenous varicose veins diagnosed in 9 target hospitals from April 2023 to August 2023, and all participants included in the trial signed an informed consent form.

Intervention

Group A: elastic bandage for 48h Group B: elastic bandage for the first 24h and then a compression full-length stocking (23-32mm Hg) for 1 week Follow-up

At baseline, patients will be asked to fill a validated visual analogue scale (VAS) , quality of life questionnaires (AVVQ), and clinical severity of varicose veins (VCSS) . They will also be asked to attend a follow-up in 1 week and at 3 months.

At 1 week, target vein closure rate will be examined by double ultrasound scan (DUS) and patients will be asked to fill VAS, AVVQ, VCSS, postoperative complications , time to return to normal work, and compliance.

At 3 months, target vein closure rate will be examined by double ultrasound scan (DUS) and patients will be asked to fill VAS, AVVQ, VCSS, postoperative complications , time to return to normal work, and compliance.

Sample Size

The target vein closure rate in the control group was set to 98%, and α=0.025 (unilateral) and (1-β)=0.9 were taken, combined with clinical expert recommendations, a non-inferiority threshold δ of -6% was taken. We would need to recruit 230 patients (115 per group) to show a difference. However, to increase the robustness of the results, considering a potential lost-to-review rate of 20% of study subjects, combined with the low probability of adverse events in this trial, the total sample size was expanded to 360.

Study duration

With 3 months follow-up, therefore, the study will be running for 12 months with a target recruitment of 360 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary unilateral lower limb saphenous varicose veins aged 18 to 80 years
2. Patients with CEAP classification of C2-C4 stage
3. 2mm≤diameter of the main trunk of the saphenous vein in the thigh segment ≤15mm
4. Agree to participate in this study and voluntarily sign the informed consent form

Exclusion Criteria:

1. Patients who have difficulty tolerating surgery
2. The main trunk of the saphenous vein is extremely twisted or tightly attached to the skin
3. Previous history of ipsilateral varicose vein surgery in the lower extremity
4. Combined deep vein thrombosis in the affected lower extremity or previous deep vein thrombosis in the affected lower extremity
5. Uncorrectable coagulation dysfunction or significant blood abnormalities with significant bleeding tendency (platelets ≤ 30*10^9/L)
6. Acute thrombosis in the saphenous vein
7. Combination of the affected lower extremity lower extremity atherosclerotic occlusive disease who
8. Ankle-brachial index ABI < 0.6 and/or absolute ankle pressure < 60 mmHg
9. Patients who cannot wear elastic stockings or are allergic to elastic bandages or elastic stockings
10. Patients during pregnancy or lactation
11. Previous history of pulmonary embolism
12. Participating in clinical trials of other drugs or devices
13. Other patients deemed unsuitable for this study by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Target vein occlusion rate as assessed by duplex ultrasound scan | 3 months post-op
  The primary outcome of the study is target vein occlusion rate at 3 months assessed with duplex ultrasound scan. Recanalisation will be defined by a segment of vein≥5cm.
  Target vein occlusion rate = Number of target venous closure cases in the group/total number of cases in the group

SECONDARY OUTCOMES:
Pain score as assessed by VAS | Baseline, 1 week post-op, 3 months post-op
  Patients will be asked to record pain scores with Visual Analogue Score (VAS)， The scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Quality of life score as assessed by AVVQ | Baseline, 1 week post-op, 3 months post-op
  Patients will be asked to fill the Aberdeen Varicose Veins Questionnaire (AVVQ) to measure health status of varicose vein patients based on symptoms and impact on daily activities. A total score ranging from 0 to 35, with 35 being worst quality of life.
Venous clinical severity score as assessed by VCSS | Baseline, 1 week post-op, 3 months post-op
  Patients will be asked to fill the Venous Clinical Severity Score (VCSS) to evaluate the severity of hallmarks of venous disease. The questionnaire consisted of ten questions, each of which was answered by 0 (none), 1 (Mild), 2(Moderate) and 3 (Severe). A total score ranging from 0 to 30, with 30 being worst quality of venous disease.
Postoperative complications | 1 week post-op, 3 months post-op
  Postoperative complications included postoperative sensory abnormalities, skin burns/discoloration, phlebitis, hematoma, infection, deep vein thrombosis, and pulmonary embolism.
Time to return to normal work | 1 week post-op, 3 months post-op
  The investigator will use a uniform question to ask the patient how long it takes to return to normal work or life, or both (days).
Compliance | 1 week post-op, 3 months post-op
  Compliance refers to the extent to which patients followed compression therapy as recommended by their clinicians.Investigators will use a uniform question to ask patients whether they have completed compression treatment as recommended by their doctors in the past week or three months.- 1 (None) , 2 (occasionally) , 3 (mostly) , and 4 (completely) . Those who did not fully follow the study protocol for compression treatment should continue to be asked about their actual compression treatment and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang Procince, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang M, Jiang W, Hong J, Li L, Shang D, Zhao Y, Liu Z, Qi M, Jin M, Zhu Y. Effect of short-term compression therapy after thermal ablation for varicose veins: study protocol for a prospective, multicenter, non-inferiority, randomized controlled trial. Trials. 2023 Oct 12;24(1):669. doi: 10.1186/s13063-023-07609-1. PMID 37828585